CLINICAL TRIAL: NCT03966989
Title: Improving Quality & Equity of Emergency Care Decisions (IQED): R21 Pilot Phase
Brief Title: Improving Quality & Equity of Emergency Care Decisions (IQED)
Acronym: IQED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to COVID-19 pandemic
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, Los Angeles (Other); Olive View-UCLA Education & Research Institute (Other); LAC+USC Medical Center (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Daniella Meeker, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-18-00522; R21AG057400 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-05-29 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Emergency Department
Keywords: Emergency Medicine; Behavioral Research
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Performance Feedback (Experimental): Feedback offline either via email or text
  Interventions: Behavioral: Performance Feedback
- Control (No Intervention): Standard practice control

INTERVENTIONS:
Behavioral: Performance Feedback — Performance feedback offline that benchmarks providers' own performance to that of their peers
  Arms: Performance Feedback

SUMMARY:
Recent work in emergency medicine has shown errors were more likely to occur at the end of shifts, as pressure exists to make a number of decisions simultaneously, and after what may be an already long series of cognitive challenges. Decision fatigue may also contribute to disparities by surfacing subconscious bias. The objective of the R21 pilot phase of Improving Quality & Equity of Emergency Care Decisions (IQED) is to identify addressable gaps in quality and equity and use performance feedback as an intervention to improve performance on chest pain, CT imaging, and antibiotic prescribing. Performance feedback intervention will include feedback offline via email or text.

DETAILED DESCRIPTION:
The objective of the R21 pilot phase of Improving Quality & Equity of Emergency Care Decisions (IQED) is to identify addressable gaps in quality and equity and use performance feedback as an intervention to improve performance on chest pain, CT imaging, and antibiotic prescribing. Performance feedback intervention will include feedback offline via email or text.

Each clinician will be randomized at the provider or clinic level to either the intervention or control group. Once clinicians are randomized, the aforementioned intervention will be turned on for a 3-6 month time period.

For providers in the intervention group, the goal is to evaluate the effect of social norms on overuse and underuse behavior related to prescriptions or testing. Near real-time social norms will be delivered to providers which benchmark their own performance on various metrics to that of their peers. The investigators performance feedback reports for each provider randomized to receive the audit and feedback intervention will have three key characteristics: (1) each target provider will receive his or her individual performance, (2) benchmarks will prominently feature the performance of providers who would be considered credible peers of the target provider, and (3) benchmarks will reflect only performance that is desirable (e.g., showing only the performance of the best-performing credible peers).

Providers randomized to the control group will follow standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Attendings and residents that see patients in the Emergency Department.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of behavioral nudges to improve quality and safety in Emergency Medicine through measurement of adherence to guidelines: Chest Pain | 6 months
  Measurement of clinician adherence to guidelines for quality measures related to chest pain (proportion of cases in which HEART score algorithm was used for chest pain patients)
Efficacy of behavioral nudges to improve quality and safety in Emergency Medicine through measurement of adherence to guidelines: CT imaging | 6 months
  Measurement of clinician adherence to guidelines for quality measures related to CT imaging (proportion of orders for unnecessary CT scans)
Efficacy of behavioral nudges to improve quality and safety in Emergency Medicine through measurement of adherence to guidelines: Antibiotic prescribing | 6 months
  Measurement of clinician adherence to guidelines for quality measures related to antibiotic prescribing (proportion of inappropriate antibiotic prescriptions for acute respiratory infections)

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Meeker, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - Lac + Usc, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Olive View Medical Center, Sylmar, California
  - Harbor UCLA, Torrance, California